CLINICAL TRIAL: NCT03374475
Title: An Exploratory, Multicenter, Placebo-controlled, Randomized, Double-blind Study to Investigate the Antidepressant Mechanism-of-action of JNJ-42847922 in Subjects With Major Depressive Disorder
Brief Title: A Study to Investigate the Antidepressant Mechanism-of-action of JNJ-42847922 in Participants With Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108382; 2017-002633-28 (EudraCT Number); 42847922MDD1009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-12-04; First posted 2017-12-15 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lead-in period: Placebo (Placebo Comparator): Participants who successfully complete the baseline examination visit at the clinical site/unit, will be treated with placebo (2 capsules taken orally) for the duration of the lead-in period which will last up to 3 weeks. Investigators and participants will be blinded to exact duration of each participant-specific lead-in period throughout the study.
  Interventions: Drug: Placebo
- Treatment period: JNJ-42847922 or Placebo (Experimental): Placebo lead-in period responders and non-responders will be randomized to receive either placebo or 20 milligram (mg) JNJ-42847922 or 40 mg JNJ-42847922 for 5 Weeks. Participants will swallow JNJ-42847922 20 mg (2*10-mg capsules) or JNJ-42847922 40 mg (2*20-mg capsules) or 2 matching placebo capsules once daily for 5 Weeks.
  Interventions: Drug: JNJ-42847922 20mg; Drug: JNJ-42847922 40mg; Drug: Placebo
- Withdrawal period: Placebo (Placebo Comparator): Participants who will complete the treatment period prior to the end of Week 8 will enter the withdrawal period where they will be treated with placebo (2 capsules taken orally) for the remaining time of the double-blind phase of the study. Investigators and participants will be blinded to exact duration of each participant-specific withdrawal period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42847922 20mg — Participants will swallow 20 mg (2*10 mg) JNJ-42847922 capsule orally for 5 weeks during treatment period.
  Arms: Treatment period: JNJ-42847922 or Placebo
Drug: JNJ-42847922 40mg — Participants will swallow 40 mg (2*20 mg) JNJ-42847922 capsule orally for 5 weeks during treatment period.
  Arms: Treatment period: JNJ-42847922 or Placebo
Drug: Placebo — All participants will receive matching placebo capsule during lead in period, treatment period and withdrawal period.

SUMMARY:
The purpose of this study is to explore if the magnitude of treatment effect (JNJ-42847922; placebo) on symptoms of depression (as measured by Hamilton rating scale for depression-17 [HDRS17], Sleep item-adjusted HDRS17, Anxiety/somatization factor score and the 6-item subscale from HDRS17 [HAM-D6]) differs across different levels of hyper-arousal status (characterized by Sleep parameters, ruminative response scale [RRS], Sleep and Worry visual analogue scale [VAS], quantitative electro-encephalography [qEEG], heart rate variability [HRV] and others).

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 35 kilogram per meter square (kg/m^2) inclusive (BMI = weight/height^2)
* Participants must be medically stable based on clinical laboratory tests, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and baseline
* Population specific: Participant must meet Diagnostic and Statistical Manual of Mental Disorders - fifth edition (DSM-5) diagnostic criteria for MDD (international classification of diseases [ICD]-code F32.x and F33.x), without psychotic features, and confirmed by the Mini International Neuropsychiatric Interview (MINI) 7.0; have a Montgomery Asberg Depression Rating Scale (MADRS) total score greater than or equal to (>=) 25 at screening and must not demonstrate a clinically significant change (that is, an improvement of greater than (>) 20 percent (%) on their MADRS total score) from the screening to the second completion of MADRS by telephone at most 4 days before the baseline visit; Not currently receiving antidepressant drug therapy for >= 2 weeks before screening
* Men who are sexually active with a women of childbearing potential (WOCBP) and have not had a vasectomy must agree to use a barrier method of birth control
* A woman of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test before the first dose
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Has failed more than 2 treatments (no more than 20 percent (%) response) with a differing pharmacological mode of action despite an adequate dose and duration during a previous, or the current depressive episode
* Has a diagnosis of Cushing's Disease, Addison's Disease, primary amenorrhea, or other evidence of significant medical disorders of the Hypothalamus pituitary adrenal (HPA) axis
* Is pregnant or breast feeding
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 60 days before the planned first dose of study drug, or has participated in 2 or more interventional clinical studies in the previous 1 year, or is currently enrolled in an interventional study
* Participant is a man who plans to father a child while enrolled in this study or within 3 months after the last dose of study drug
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Hamilton Rating Scale for Depression-17 (HDRS17) Total Score | Baseline up to Day 57
  The HDRS17 is a Clinician-Administered rating scale designed to assess the severity of symptoms in participants diagnosed with depression with a total score range of 0 to 52. It is the most widely used symptom severity measure for depression. Each of the 17 items is rated by the clinician on either a 3- point (0 to 2) or a 5-point scale (0 to 4). The point scale uses a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). Total score will be calculated by summing up the individual item score. The higher the score, the more severe the depression.
Change From Baseline in Hamilton Rating Scale for Depression-17 (HDRS17) Sleep Item-Adjusted Total Score | Baseline up to Day 57
  The HDRS17 is a Clinician-Administered rating scale designed to assess the severity of symptoms in participants diagnosed with depression with a score range of 0 to 52. It is the most widely used symptom severity measure for depression. Each of the 17 items is rated by the clinician on either a 3- point (0 to 2) or a 5-point scale (0 to 4). The point scale uses a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). Higher scores indicate worsening. HDRS17 Sleep Item-Adjusted is derived from the HDRS17 scale excluding the 3 sleep items (4, 5, and 6) from the total score.
Change From Baseline in Hamilton Rating Scale for Depression-17 (HDRS17) Anxiety/Somatization Factor Score | Baseline up to Day 57
  The HDRS17 anxiety/somatization factor derived from Cleary and Guy's factor analysis of the HDRS scale, includes six items from the original 17-item version: the items for psychic anxiety, somatic anxiety, gastrointestinal somatic symptoms, general somatic symptoms, hypochondriasis, and insight. Anxious depression is often defined as Major Depressive Disorder (MDD) with high levels of anxiety symptoms, as reflected in an anxiety/ somatization factor score greater than or equal to (>=) 7. The score ranges from 0 to 18, with higher scores indicating greater severity of symptoms.
Change From Baseline in 6 Item Subscale From HDRS17 (HAM-D6) Score | Baseline up to Day 57
  The 6-Item Hamilton Depression Scale (HAMD-6), derived by the sum of HAMD-17 items (the six items in the HAM-D6 are: depressed mood, guilt feelings, work and interests, psychomotor retardation, psychic anxiety, and general somatics [tiredness and pains]), evaluates "core" symptoms of Major Depressive Disorder (MDD). Total subscale scores range from 0 (normal) to 22 (severe). The higher the score, the more severe the depression.

SECONDARY OUTCOMES:
Change From Baseline in Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR16) | Baseline up to Day 67
  The QIDS-SR16 is a patient reported measure designed to assess the severity of depressive symptoms. The total score ranges from 0 to 27. Using a scale of severity of depression of none, mild, moderate, severe, and very severe, corresponding QIDS-SR16 total scores are none 1 to 5, mild 6 to 10, moderate 11 to 15, severe 16 to 20 and very severe 21 to 27.
Association Between Major Depressive Disorder (MDD) Symptoms and Signals of Hyper-Arousal | Baseline up to Day 67
  Association between major depressive disorder (MDD) symptoms and signals of hyper-arousal (as measured by electro-encephalography [EEG], polysomnography, and/or measures of autonomic arousal - heart rate variability) will be assessed by means of correlation analysis and mixed effect models.
Performance Score on a Cognitive Test Battery Evaluated by Symbol Digit Matching Test (SDMaT) | Baseline
  The SDMaT measures the time to pair abstract symbols with specific numbers. The test includes a coding key consisting of 9 abstract symbols, each paired with a number ranging from 1 to 9. Following the key, the participant is presented with randomly ordered symbols and is required to respond orally by naming the number or enter the number corresponding to each symbol as fast as possible using a keypad. The number of correct substitutions within 90 seconds is recorded by computerized cognitive test battery.
Performance Score on a Cognitive Test Battery Evaluated by Word List Recall Test (WLRT) | Baseline
  The WLRT used for the computerized test battery that measures person's ability to encode, consolidate, store, and retrieve verbal information and is a sensitive test of verbal learning and memory in a variety of disease states, including MDD. The memory test will include a list of 15 words presented aloud, one at a time, through the iPad. After the 15-word list is presented, the participant will be asked to verbally recall as many of the words as possible. The 15 word list and participant recall will be conducted 4 more times (total 5 times). After the 5th learning trial and recall, performance on the learning trials of the original word list and on the delayed recall will be considered as the primary scores. The computer tablet will record and score the participant's responses to the evaluation.
Performance Score on a Cognitive Test Battery Evaluated by Trail Making Test Form B (TMT-B) | Baseline
  The computerized (Revere.D) version of the TMT-B is modeled after the paper-and-pencil version of the test. The TMT-B measures divided attention and executive function (tracking and sequencing). The participant is instructed to draw a line to connect a set of 25 consecutively numbered and lettered circles, alternating sequentially between numbers and letters (that is, 1 A 2 B). The participant is instructed to work as quickly as possible while still maintaining accuracy. The TMT-B has acceptable reliability; reliability coefficients have typically been reported as exceeding 0.65. The TMT-B is sensitive to cognitive decline associated with MDD.
Change From Baseline in Bond & Lader (B&L) Visual Analogue Scale (VAS) | Baseline up to Day 57
  The B&L VAS is made up of 16 pairs of alternative descriptors of mood and attention at either end. The Bond-Lader of a 10 cm line. Participants will rate their feelings at the time of assessment by indicating the point on the line which best represent their mood. Each item is scored by measuring the position relative to the left hand end of the line and levels of anxiety, sedation, and dysphoria are then calculated from the combined scores of selected items. The score ranges from 0 to 100, with a high score reflecting a high level of anxiety, sedation or dysphoria.
Change From Baseline in Profile of Mood States (POMS) | Baseline up to Day 57
  The POMS measures individuals' mood states. The POMS measures individuals' mood states. This is a validated scale to measure positive and negative mood states. The POMS contains 30 items and assesses six identified mood factors: Tension-Anxiety, Depression-Ejection, Anger- Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. Scoring of the instrument provides a global score of 0 to 120 or individual domain scores. Lower scores indicate better mood state. The POMS brief form is a simple self-rating instrument.
Plasma Concentration of JNJ- 42847922 and its Metabolites | Day 36 to 40 (over 48 hours during Visit 6)
  Plasma concentration assessment will be done to characterize the pharmacokinetics (PK) of JNJ-42847922 and its metabolites.
Percent Change From Baseline in Biomarker Levels | Day 36 to 40 (over 48 hours during Visit 6)
  Percent change from baseline in biomarker includes high-sensitivity (hs) C-reactive protein (CRP), interleukin(IL) 6, IL10, IL1b, tumor necrosis factor (TNF) alpha, cortisol, growth hormone, adiponectin, leptin, brain-derived neurotrophic factor (BDNF), Insulin-like growth factor 1 (IGF1), interleukin-6 receptor (IL6R), insulin, glucose, adrenocorticotropic hormone, Kynurenine metabolites will be assessed.
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to end of the study (Day 67)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (14):
- United States (3):
  - Artemis Institute for Clinical Research, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Qps-Mra, Llc, Miami, Florida
- Belgium (2):
  - SGS Phase 1 Unit AZ St-Maarten, Mechelen
  - Clinical Pharmacology Unit, Merksem
- Germany (4):
  - Charite Research Organisation GmbH, Berlin
  - Emovis GmbH, Berlin
  - Fraunhofer-Institut für Toxikologie und Experimentelle Medizin, Hanover
  - Somni Bene GmbH, Schwerin
- Centre for Human Drug Research, Leiden, Netherlands
- United Kingdom (4):
  - MAC Clinical Research, Blackpool
  - MAC Clinical Research, Liverpool
  - Hammersmith Medicines Research, London
  - MAC Clinical Research, Manchester

REFERENCES:
- [Derived] Mesens S, Kezic I, Van Der Ark P, Etropolski M, Pandina G, Benes H, Savitz A, Drevets WC. Treatment effect and safety of seltorexant as monotherapy for patients with major depressive disorder: a randomized, placebo-controlled clinical trial. Mol Psychiatry. 2025 Jun;30(6):2427-2435. doi: 10.1038/s41380-024-02846-5. Epub 2024 Dec 11. PMID 39663378